CLINICAL TRIAL: NCT06170619
Title: A Prospective, Post-Approval, Open-Label, Multi-Center United States (US) Registry to Evaluate the Effectiveness and Safety of Obsidio in Clinical Practice
Brief Title: Obsidio™ Conformable Embolic Registry
Acronym: OCCLUDE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2513
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hypervascular Tumors; Bleeding; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All subjects
  Interventions: Device: Obsidio™ Conformable Embolic

INTERVENTIONS:
Device: Obsidio™ Conformable Embolic — Embolization with Obsidio™ Conformable Embolic.

SUMMARY:
OCCLUDE is a prospective, post-approval, open-label, single arm, multi-center US registry of patients who undergo embolization with Obsidio™ Conformable Embolic. The purpose of this Registry is to assess effectiveness and safety outcomes of subjects who undergo embolization with Obsidio.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age
* Signed informed consent*
* Patient is to undergo or has undergone embolization with Obsidio™ Conformable Embolic
* Patient is willing and able to comply with protocol requirements, including all procedures, clinical evaluations, and follow-up visits *Patients being treated for control of bleeding/hemorrhage who are unable to consent prior to their procedure, can be enrolled if the informed consent is provided and signed within 72 hours of the index procedure

Exclusion Criteria:

* Patient has a life expectancy < 30 days
* Contraindications to receiving Obsidio™ Conformable Embolic per the Instructions For Use (IFU)
* Embolization for uterine fibroids, prostate artery, genicular artery, ovarian vein, spermatic vein, pulmonary arteriovenous malformations, bronchial artery, asymptomatic benign tumors, portal vein, varices, lymphatic/thoracic duct, nonvascular channel (e.g. ureter, intestinal fistula)
* Patients with more than 2 discrete lesions, defined as a treatment area that may be fed by one or more vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo or have undergone embolization with Obsidio™ Conformable Embolic
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness endpoint | Immediately following index procedure
  The primary effectiveness endpoint is technical success, which is defined as occlusion of the target vessel(s) after embolization with Obsidio™ Conformable Embolic as assessed via angiography or demonstration of a cast of Obsidio occluding the artery on fluoroscopy or image acquisition immediately following the index procedure.
Primary safety endpoint | 30 days following index procedure
  The primary safety endpoint is freedom from major adverse events defined as non-target embolization events that meet serious adverse event criteria, unintended target organ or soft tissue infarction, vessel perforation/injury and catheter entrapment through 30 days of the index procedure.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - St. Joseph's Medical Center, Stockton, California
  - Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mercy Hospital, Coon Rapids, Minnesota
  - Barnes Jewish Hosital, St Louis, Missouri
  - University Hospital, Newark, New Jersey
  - Albany Medical Center, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Houston Health Science Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No